CLINICAL TRIAL: NCT05990959
Title: Risk Factors, Prognosis, and Potential Chemoprevention Drugs in Patients With Recurrent Hepatocellular Carcinoma After Curative Surgeries: a Nationwide Retrospective Cohort Study and a Multi-center Prospective Cohort Analysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Collaborators: Ministry of Health and Welfare, Taiwan (Other Government)
Responsible Party: Principal Investigator, Chun Chieh Yeh, Dr., China Medical University Hospital
Other Study IDs: CMUH111-REC2-039
Record Dates: First submitted 2023-08-05; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Hepatocellular Carcinoma Recurrent; Surgery
Keywords: hepatocellular carcinoma; Recurrent; Surgery; Chemoprevention; National Health Insurance Research Database
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Biospecimen would be retrieved from already stored biobank in our own affiliation .The biospecimen may contain blood and liver tumors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HCC_surg: HCC surgical patients who would receive surgical interventions based on clinical judgment and would donate biospecimen for research after signing informed consent permission.
  Interventions: Other: No intervention for research purpose

INTERVENTIONS:
Other: No intervention for research purpose — No any intervention will be applied under research purpose. All procedure or drugs would be given to the patient under best clinical judgment, not for research purpose.

SUMMARY:
Backgrounds: Surgeries are the mainstream of curative therapies for hepatocellular carcinoma (HCC). However, high risk of recurrent HCC after liver surgeries is still the unsolved clinical issue (early recurrence 21% per year; late recurrence 18% per year). Early recurrence mainly result from disseminated HCC; by contrast, late recurrence usually originate from carcinogenic microenvironment. Currently, no large-scale nationwide studies that integrate laboratory date and clinical information was performed to investigate risk factors and prognosis of post-operative recurrent HCC. Besides, owing to economic issue, few companies would initiate pharmacologic studies to investigate chemoprevention agents for HCC. Furthermore, few biomarkers were discovered from Taiwanese HCC cohort to predict post-operative tumor recurrence because of no standardized cooperative platforms to share biological tissue and clinical information. Therefore, we wish to utilize a nationwide retrospective cohort from integrated national health insurance database (NHIRD) and a prospective multi-center clinical cohort study to address aforementioned issues.

Aims:

1. Investigate risk factors and prognosis of post-operative recurrent HCC in Taiwanese cohort
2. Discover chemoprevention targets from generic drugs to reduce risk of post-operative recurrent HCC
3. Determine biomarkers from Taiwanese cohort in prediction of post-operative recurrent HCC

DETAILED DESCRIPTION:
Study subject and methods:

Nationwide retrospective cohort study

1. Establish prediction models for postoperative recurrent HCC by analyzing surgical HCC patients' clinical information and perioperative laboratory date based on the database of a nationwide retrospective cohort organized by the Ministry of Health and Welfare and Health insurance office
2. Discover chemoprevention agents in association with reduced risk of post-operative recurrent HCC using the aforementioned database

Multicenter prospective cohort study:

1. To discover biomarkers in prediction of post-operative recurrent HCC , we will establish a shared platform to prospectively and systemically collect Taiwanese HCC surgical patients' bio-materials and clinical information from China Medical University Hospital, Asian University Hospital, Mackay Hospital, Taichung Veterans General Hospital, E-Da Hospital,…etc.
2. Using the multicenter prospective cohort, we could validate the results from the nationwide retrospective cohort study, and even improve the prediction models by adding biological parameters that are not available in the nationwide retrospective cohort

Hospital biobank based retrospective case-control study Investigate clinical and biological parameters in prediction of tumor recurrence in HCC surgical patients by hospital based biobank and relevant clinical information

Laboratory in-vivo and in-vitro study Investigate causal relationship between prognosis of HCC and selected biomarkers from above studies as well as four universal tumor theragnostic markers (ADAM9, MTHFD2, RRM2, and SLC2A1) and explore treatment effects of corresponding inhibitors

Expected results: For scientists, they may benefit from the shared database of Taiwanese HCC surgical patients for the HCC related researches; for physicians, they could predict risk of post-operative recurrent HCC in Taiwanese HCC patients and use generic drugs as potentially chemopreventive drugs for HCC; for patients, they could benefit from the personalized medical advice to increase the survival; for the authorities, they could design a policy to reduce the risk of post-operative recurrent HCC, and even prolong HCC patients' survival in a cost-effective way by using generic drugs as chemopreventive regimens for HCC.

ELIGIBILITY:
Inclusion Criteria:

* All HCC surgical patients aged more than 20 year-old who sign informed consent for donating remnant tissue or blood after liver surgeries

Exclusion Criteria:

* Pregnant women

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All HCC surgical patients aged more than 20 year-old who sign informed consent for donating remnant tissue or blood after liver surgeries that would be performed under best clinical judgment, NOT for research purpose.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 year
  Overall survival
Disease free survival | 5 year
  Disease free survival

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Chieh Yeh, Dr., Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Department of Surgery, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No
All patient's privacy would be protected under our IRB regulation. Thus, I cannot release IPD.